CLINICAL TRIAL: NCT05704556
Title: A Phase 1, Open-label Study to Evaluate the Pharmacokinetics and Safety of Single Doses of VX-548 in Subjects With Severe or Moderate Renal Impairment and in Matched Healthy Subjects
Brief Title: Evaluation of the Pharmacokinetics and Safety of VX-548 in Participants With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX22-548-014
Record Dates: First submitted 2023-01-19; First posted 2023-01-30 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Cohort 1: Severe Renal Impairment (Experimental): Participants will receive a single dose of VX-548 in a fasted state.
  Interventions: Drug: VX-548
- Cohort 2: Matched Healthy Participants (Experimental): Healthy participants matched to cohort 1 will receive a single doses of VX-548 in a fasted state.
  Interventions: Drug: VX-548
- Cohort 3: Moderate Renal Impairment (Experimental): Participants will receive a single dose of VX-548 in a fasted state.
  Interventions: Drug: VX-548
- Cohort 4: Matched Healthy Participants (Experimental): Healthy participants matched to cohort 3 will receive a single dose of VX-548 in a fasted state.
  Interventions: Drug: VX-548

INTERVENTIONS:
Drug: VX-548 — Tablets for oral administration.
  Other Names: Suzetrigine

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (PK), safety, and tolerability of VX-548 and its metabolite in participants with severe or moderate renal impairment and healthy participants.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4) (A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Cohorts 1 and 3: Participants with Severe or Moderate Renal Impairment

  * Body mass index (BMI) of greater than or equal to (>=)18.0 to less than (<) 40.0 kilogram per square meter (kg/m^2)
  * Stable renal function as pre-defined in the protocol
* Cohorts 2 and 4: Matched Healthy Participants

  * Healthy participants will be matched to Cohorts 1 and 3 participants according to each of the following parameters: sex, age (±10 years), and BMI (±15%)

Key Exclusion Criteria:

* Cohorts 1 and 3: Participants with Severe or Moderate Renal Impairment

  * Hemoglobin less than or equal to (≤) 9.0 gram per deciliter (g/dL) at screening
* Cohorts 2 and 4: Matched Healthy Participants

  * Prior renal transplantation, prior hemodialysis, or prior peritoneal dialysis
* All Cohorts:

  * History of febrile or acute illness that has not fully resolved by 14 days before study drug dosing.
  * Any condition possibly affecting drug absorption

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of VX-548 and its Metabolite | Day 1 to Day 14
Area Under the Plasma Concentration Versus Time Curve From the Time of Dosing Extrapolated to Infinity (AUC0-inf) of VX-548 and its Metabolite | Day 1 to Day 14

SECONDARY OUTCOMES:
Apparent Clearance of VX-548 | Day 1 to Day 14
Apparent Renal Clearance of VX-548 and its Metabolite (CLr) | Day 1 to Day 14
Apparent Non-Renal Clearance of VX-548 | Day 1 to Day 14
Safety and Tolerability as Assessed by Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Day 1 to Day 23
Fraction Unbound (fu) for VX-548 and its Metabolite in Plasma | Day 1 to Day 2
Unbound Area Under the Concentration Versus Time Curve of VX-548 and its Metabolite | Day 1 to Day 14

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Infigo Clinical Research, DeLand, Florida
  - Clinical Pharmacology of Miami, LLC, Miami, Florida
  - GCP Research, St. Petersburg, Florida
  - Genesis Clinical Research, Tampa, Florida
  - Elixia, Phase 1 Clinical Site, Tampa, Florida
  - Southwest Houston Research, Ltd, Houston, Texas
  - Clinical Trials of Texas, LLC, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing